CLINICAL TRIAL: NCT05657509
Title: Effects of Functional Training on Physical Fitness, Hockey Skills and Functional Movement Among Elite Male Field Hockey Players in Pakistan
Brief Title: Effects of Functional Training on Field Hockey Players Physical Fitness, Hockey Skills and Functional Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Marrium Bashir, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: GS61096
Record Dates: First submitted 2022-11-18; First posted 2022-12-20 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Physical Inactivity
Keywords: Physical fitness components; Hockey skills; Functional movement screen
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group will continue functional training exercises and the control group will exercise traditional type with coaches' guidelines. Each group has equally male players.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male field hockey players of Functional training (Experimental): Functional training exercises focus on improving physical fitness and movement skills performance. Functional training targets the neuromuscular system through engagements of muscle groups as well as nerve function to optimize movements. The present study applied functional training to elite male field hockey players to assess fitness level as well as skill performance. Post-test 1 will be after 6 weeks, and post-test 2 after 12 weeks to measure performance.
  Interventions: Other: Functional training
- Male field hockey players of traditional regular type of training exercises (Active Comparator): The traditional training method involves exercises to increase the strength and durability of a certain muscle. Male field hockey players will be continuing their regular traditional type training exercises for 12 weeks.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Functional training — Functional training Length: 12 weeks; Training duration: 60 minutes; Intensity: 60 to 95%; 3 days per week. The intensity of the training is increasing in the first 20 minutes, and the intensity is gradually decreasing in the next 5 minutes; Rest: 30 seconds rest between exercises and 1-2 minute rest between sets.
  Arms: Male field hockey players of Functional training
Other: No intervention — The Control group continues regular traditional training exercises for 12 weeks with a training duration of 60 minutes and three days per week.
  Arms: Male field hockey players of traditional regular type of training exercises

SUMMARY:
Functional training is an exercise modality that emphasizes functional, multi-joint movements that can be modified to any fitness level and elicit greater muscle recruitment. This training refers to an exercise program that is characterized by relatively short bursts of vigorous activity, interspersed by periods of rest or low-intensity exercise for recovery. Even though this type of training has been used among athletes since the later part of the 20th century, it recently has gained momentum among fitness enthusiasts and has been identified as a "Top 10 Fitness Trend" in 2018. However, recent work shows that the magnitude of these effects on body structures and functions may be rather modest in nature with potentially differing directions. Furthermore, players' ability to create actions at a very fast pace has a significant impact on the course and result of the game. Finally, to evaluate that functional training can improve male field hockey players' physical fitness, hockey skill and functional movements.

DETAILED DESCRIPTION:
This study included two groups, namely the control and functional training groups. The sample is 19-23-year-old Pakistani elite male hockey players who do not do functional training exercises. Based on the literature review, the training frequency of this experiment was arranged three (3) times/week, the total training duration will be 12 weeks, and the time of each training session will be changed over two weeks. The 12 weeks of exercise last 60 minutes, excluding 10-minute warm-up and a 10-minute cool-down. Training intensity ranges from 60 to 95%. Teach all sports techniques before the intervention. In contrast, the control group discussed with their coaches and will continue the 12-week traditional type of regular exercise.

Content of Experimental Group: Week 1-2: Introduces the classification of Functional training, starting from the plank and movement exercises; Week 3-4: exercises to improve physical fitness lateral bridging with alternating leg, flexion and leg extension exercises ; 5-6 Week : Reviewed the basic hockey skills, introduced the exercises, high knee run drill, two-foot lateral hops in and out basic step, One lower limb up and side plank, Incline push-ups, Lateral pull-up, feet on Swissball, Straddle squat hops; 7-8 Week: Learn the exercises, jumping jack variations drill, diamond push up, medicine ball rebound lateral toss, prone press up wall sit bilateral reach, icky Shuffle, Crunches; 9-10 Week: Review the lateral bridging with hip abduction (90 knee angle), cross limbs up and one leg up side plank, active leg lowering to bolster, Prone kneeling, Double step icky shuffle, 5-10-5 cone agility drills; 11-12 Week: Review physical fitness, hockey skills and functional movement screening, exercises with medicine ball curl up chest, lateral hope explosive medicine ball, One arm push-up with Swiss ball, clapping push-ups, standing pull ups, Squats chops, 5-10-5 cone agility drills.

ELIGIBILITY:
Inclusion Criteria:

* The population must be elite male hockey players between the ages of 19 to 23
* Able to perform all tests and be Physically active (no previous experience performing functional training)
* Only players who understand the study purposes and procedures and can complete this training requirement can be included in the research data

Exclusion Criteria:

* Female field hockey players should be excluded from this study
* On medication that may affect body composition and muscles activity
* Presently engaged in regular functional training programs
* Players who are consistently late or absent from training sessions will eventually be excluded

Ages: 19 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Speed performance of field hockey players | 2 weeks
  30-meter sprint test use to monitor the speed of the individual. Previous research demonstrated that the 20m sprint test measurement also has a high reliability.
Agility performance of field hockey players | 3 weeks
  The Illinois Agility measure the participants agility. Then participants sprinted up to the second 10-meter cone, turned around, and made their way back to the finish cone. The best time of two attempts will be recorded. Previous research demonstrated that the Illinois Agility test measurement also has a high reliability value 0.96 (95% CI, 0.85 - 0.98).
Flexibility of field hockey players | 4 weeks
  Flexibility will be assessed through Sit and Reach test. The maximal reach distance will record in centimeters for all 3 trials. The purpose of this test is to assess the flexibility of the lower back and hamstring. Previous research showed the intra-class correlation coefficient for test-retest reliability for the sit and reach test was 0.93.
Muscular strength of field hockey players | 6 weeks
  Muscular strength will be assessed through 1RM test. According to the previous studies test-retest ICCs ranged from 0.64 to 0.99 (median ICC = 0.97), where 92% of ICCs were ≥ 0.90, and 97% of ICCs were ≥ 0.80. It can be concluded that the 1RM test generally has good to excellent test-retest reliability, part of the body assessed (upper vs. lower body) of participants.
Functional movement screen of field hockey players | 8 weeks
  Functional movement screen using the standard 0-3 ordinal system. A score of 3 will be given for performing the specific movement perfectly, a 2 given when the movement complete with some compensatory movements observe, a score of 1 given when the subject could not complete the movement, and a score of 0 associate with pain being present during the movement. Functional movement assesses through the FMS Kit.
Dribbling skill performance of field hockey players | 10 weeks
  The slalom sprint and dribble test will be use as the criterion standard for measuring construct validity. Previous research demonstrated that the test-retest reliability (ICC) of the single-task dribble test is 0.78; suggesting that this is a reliable test.
Shooting skill performance of field hockey players | 12 weeks
  Shooting accuracy valuate by placing a hockey ball at five positions in the goal scoring area ("D"). This test will carry out within the goal area. Each player had eight shots executed from five different positions, previously established, in the direction of the goal; four shots were hit from positions 1 to 4, two were pushed from positions 2 and 3, and two flick shots were taken from position 5. Each shot made was given 1 point, and failed shots were given 0, ranging from 0 to 8 points.

CONTACTS AND LOCATIONS:
Overall Officials: Marrium Bashir, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Hockey training center, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Yildiz S, Pinar S, Gelen E. Effects of 8-Week Functional vs. Traditional Training on Athletic Performance and Functional Movement on Prepubertal Tennis Players. J Strength Cond Res. 2019 Mar;33(3):651-661. doi: 10.1519/JSC.0000000000002956. PMID 30431536
- [Background] Sander A, Keiner M, Schlumberger A, Wirth K, Schmidtbleicher D. Effects of functional exercises in the warm-up on sprint performances. J Strength Cond Res. 2013 Apr;27(4):995-1001. doi: 10.1519/JSC.0b013e318260ec5e. PMID 22692105
- [Background] Keiner M, Kadlubowski B, Sander A, Hartmann H, Wirth K. Effects of 10 Months of Speed, Functional, and Traditional Strength Training on Strength, Linear Sprint, Change of Direction, and Jump Performance in Trained Adolescent Soccer Players. J Strength Cond Res. 2022 Aug 1;36(8):2236-2246. doi: 10.1519/JSC.0000000000003807. Epub 2020 Aug 27. PMID 32868678
- [Background] Baron J, Bieniec A, Swinarew AS, Gabrys T, Stanula A. Effect of 12-Week Functional Training Intervention on the Speed of Young Footballers. Int J Environ Res Public Health. 2019 Dec 24;17(1):160. doi: 10.3390/ijerph17010160. PMID 31878326